CLINICAL TRIAL: NCT05444270
Title: Prospective Multi-institutional Phase III Trial of Salvage Systemic Therapy With or Without Stereotactic Ablative Radiotherapy for Recurrent Ovarian Cancer
Brief Title: Salvage Systemic Therapy With or Without Stereotactic Ablative Radiotherapy for Recurrent Ovarian Cancer
Acronym: SABR-ROC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2022-0286
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Recurrent Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard salvage therapy (Active Comparator): Subjects will continue to receive current salvage treatment suitable for subjects at the discretion of their doctor, considering the location and size of recurrence, and the patient's comorbidities.
  Interventions: Other: Standard salvage therapy
- Standard salvage therapy + SABR (Experimental): Subjects receive SABR for lesions found in imaging studies. Before or After SABR, standard salvage treatment continues as planned at the discretion of the doctor.
  Interventions: Radiation: Standard salvage therapy + SABR

INTERVENTIONS:
Other: Standard salvage therapy — Subjects will continue to receive current salvage treatment suitable for subjects at the discretion of their doctor, considering the location and size of recurrence, and the patient's comorbidities.
  Arms: Standard salvage therapy
Radiation: Standard salvage therapy + SABR — Subjects receive SABR for lesions found in imaging studies. Before or After SABR, standard salvage treatment continues as planned at the discretion of the doctor.
  Arms: Standard salvage therapy + SABR

SUMMARY:
Rationale Ovarian cancer is the 3rd most common gynecologic malignancy in Korea. The standard treatment is tumor debulking surgery with or without adjuvant chemotherapy. However, with a recurrence rate of 80%, the treatment results are the worst among gynecological cancers. The use of target and immune agents have demonstrated to improve survival. However, long-term maintenance of systemic therapy is often difficult because recurrent tumors do not respond uniformly to systemic therapy.

In the 1980~1990s, whole abdomen irradiation had been tried and faded out owing to many side effects with the introduction of taxane. Efforts have been made to find the role of salvage radiation therapy (RT) in recurrent ovarian cancer. Involved field radiotherapy (IFRT) emerged to cover the gross tumor plus regional microscopic disease in addition to salvage chemotherapy. It showed high local control, provided chemotherapy holiday in selected cases, but did not prevent out-field progression. Stereotactic ABlative Radiotherapy (SABR) is the latest treatment using an intensity modulated technique to increase the fractional dose, reduces the number of treatments, and destroys the tumor with high accuracy. SABR-COMET study, a representative clinical study, showed a significant increase in overall survival in solid cancers.

Objectives The primary objective; to evaluate whether the addition of SABR to standard salvage treatment significantly improves 3-year overall survival (OS) in patients with recurrent ovarian cancer.

The secondary objectives;

* to check whether it significantly affects quality of life (Health-related QoL), patient-reported outcome (PRO)
* to develop an deep learning-based predictive model for the treatment response of ovarian cancer subjects using radiomic and genomic analysis.

Study design Arm 1; Standard salvage therapy Subjects will continue to receive current salvage treatment suitable for subjects at the discretion of their doctor, considering the location and size of recurrence, and the patient's comorbidities.

Arm 2; Standard salvage therapy+ SABR Subjects receive SABR for lesions found in imaging studies. Before or After SABR, standard salvage treatment continues as planned at the discretion of the doctor.

Stratification factors

1. The number of No ascites, Platinum-sensitive, Normal CA125 and ECOG０-１; 0~3 vs. 4
2. Location of the lesion; Lymph node lesion vs. Non-lymph node lesion
3. PARP inhibitor; Used vs. Not used

Randomization Arm 1 : Arm 2 = 1 : 2

Estimated Accrual :

* The sample size 270 was calculated by setting the sample size to a Type I error rate (α) of 0.05 and Statistical Power of 80% using 2-Sided Equity and log-rank test.
* Accurate time: 2 years, Follow-up: 3 years (total 5 years)
* Alpha = 0.05, Power = 80%
* 1 year drop-out: 5% per group
* 3 year survival proportion: RT group 74.42%, No RT group 58%
* Arm 1: Arm 2 = 1 : 2 ratio

DETAILED DESCRIPTION:
Treatment Plan Arm 2; SABR Number of Fractions Preferred Doses Acceptable Doses

1 20 Gy 16-24 Gy 3 30 Gy 24-33 Gy 5 35 Gy 25-40 Gy 10 40 Gy 35-45 Gy

Patient Evaluation:

* Interviews
* It was performed 3, 6, 9, 12, 18, 24, 30, and 36 months after the end of treatment.
* Medical history listening, physical examination and assessment of all possible side effects
* The relevant examination can be prescribed if necessary.
* Imaging examination
* one of CT or PET-CT including areas suspected of recurrence or treatment is possible.
* If PET-CT was not performed within two months before treatment, it is recommended to perform PET-CT before treatment NOTE: Before treatment, it is recommended to perform the same examination as the imaging test that evaluated the treatment site.
* Tumor marker CA125 examination: performed on every visit after radiation therapy.
* Survey EORTC-QLQ-C30 questionnaire; prior to radiation therapy, 12, 24, and 36 months after treatment FACIT-TS-G (Arm 2 subjects); before radiation therapy, 12, 24, and 36 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed epithelial ovarian cancer
* Should have completed standard treatment for the primary tumor initially. (In the case of advanced ovarian cancer, maximal debulking operation and adjuvant platinum-based chemotherapy are performed according to the stage)
* Number of metastases allowed: ≤ 10 (Adjacent lesions can be counted as a single lesion if possible to be included in a single radiotherapy treatment plan) (left cervical lymph node, right cervical lymph node, center of the left lung, periphery of the left lung, left pleura, center of the right lung, periphery of the right lung, right pleura, mediastinal lymph node, left lobe of the liver, right lobe of the liver, perihepatic space, spleen, perisplenic space, within 2 vertebrae above or below based on the spine with the lesion, abdominal cavity, pelvic cavity, paraaortic lymph node, and pelvic lymph nodes)
* Maximum diameter of each metastasis site of gross tumor ≤ 5 cm
* Age ≥ 19 year old
* Sufficient bone marrow function on tests performed within 60 days prior to study enrollment, including:

  * Absolute neutrophil count (ANC) ≥ 500 / mm3
  * Platelet ≥ 50,000 / mm3
  * Hb ≥ 8.0 g / dl (Treatments such as blood transfusions to maintain hemoglobin count are permitted)
* Zubrod daily living performance ≤ 2 within 60 days prior to study enrollment
* Subjects must submit research-related informed consent prior to participation in the study

Exclusion Criteria:

* Brain metastasis
* Diffuse peritoneal carcinomatosis
* Exudative, hematological, or cytologically proven malignant exudate (Malignant pleural effusion)
* If previously treated with radiation therapy to metastases
* When targeting is difficult because the boundary of the metastasis site is not clear
* Coexisting or previous invasive cancer (excluding Thyroid cancer, Cervix CIS, basal cell carcinoma of skin, early gastric cancer) has not been disease-free for more than 3 years.
* Pregnancy
* Serious comorbidities defined as below

  * Unstable angina or congestive heart failure requiring hospitalization within the last 6 months
  * Deep myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of enrollment
  * At the time of enrollment, exacerbation of chronic obstructive pulmonary disease or other respiratory disease that requires hospitalization or makes it difficult to proceed with treatment in this study.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 270 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
overall survival (OS) | 3year
  to evaluate whether the addition of SABR to standard salvage treatment significantly improves 3-year overall survival (OS) in patients with recurrent ovarian cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park S, Kim H, Wee CW, Kim YS, Choi JH, Kim YS, Lee JH, Choi Y, Kim JH, Cho Y, Kim HJ, Park YJ, Park W, Eom KY, Kim YH, Kim YB. Radiotherapy quality assurance program of ongoing clinical trial using stereotactic ablative radiation therapy for recurrent ovarian cancer (SABR-ROC): a dummy run study of a prospective, randomized, multicenter phase III trial (KGOG 3064/KROG 2204). BMC Cancer. 2025 Aug 18;25(1):1336. doi: 10.1186/s12885-025-13892-9. PMID 40826041
- [Derived] Kim YB, Byun HK, Wee CW, Kim H, Kim S, Yang G, Kim J, Park SJ, Lee JY. Study protocol for prospective multi-institutional phase III trial of standard of care therapy with or without stereotactic ablative radiation therapy for recurrent ovarian cancer (SABR-ROC). BMC Cancer. 2023 Oct 20;23(1):1014. doi: 10.1186/s12885-023-11407-y. PMID 37864152